CLINICAL TRIAL: NCT05561166
Title: Study of the Determinants of Dream Recall and Content in Patients With Epilepsy
Brief Title: EPIDREAM 1 : Study of Dreaming in Epilepsy
Acronym: EPIDREAM 1
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL22_0745
Record Dates: First submitted 2022-09-27; First posted 2022-09-30 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2023-01

CONDITIONS: Epilepsy
Keywords: Epilepsy; Dreams; Seizures
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: EPIDREAM Questionnaire — EPIDREAM Questionnaire (questionnaire about dreams and epileptic seizures)

SUMMARY:
Dreaming is a sleep-associated cognitive process whose neural substrates and functions remain poorly understood. In healthy subjects, the frequency of dream recall is influenced by several factors such as age, gender, interest in dreams and sleep quality. The content of dreams mainly depends on waking life experiences, especially when they are recent and have a strong emotional content. The function of dreams remains debated but it is widely accepted that dreams play a role in emotional regulation.

Modifications in dreams are observed in several neurological diseases and sleep disorders, due to the modifications of sleep related to these diseases, as well as to associated disturbances in cognitive functioning and to the impact on such diseases on waking life. Epilepsy is a neurological condition characterized by a predisposition to seizures resulting from excessive and synchronized abnormal brain activity; it is associated with numerous co-morbidities including sleep and cognitive disorders, which are present in nearly one in two patients. However, the influence of epilepsy on sleep-related cognitive processes is poorly understood. It is suspected that nocturnal epileptic activity disturbs sleep-related memory consolidation processes, but the consequences of epilepsy on dreams have been little investigated.

The study of the determinants (epilepsy syndrome, location of the epileptic focus, presence of sleep-related seizures, certain anti-epileptic treatments, alteration of the quality of sleep) of dream characteristics in this context could lead to a better understanding of the dreams physiology, the interactions between epilepsy and sleep, as well as the cognitive and emotional functioning related to sleep in epilepsy. It could also determine whether dream characteristics can provide information on the epilepsy syndrome and on the presence of nocturnal seizures, and thus constitute a diagnostic tool.

In this cross-sectional observational study, we aim to identify determinants of dream recall in relation to epilepsy by administering a simple and brief questionnaire on sleep and dreams, to all consecutive patients seen in epileptology consultation during 12 months. Our objectives are

1. To determine whether the presence of sleep-related seizures influences the frequency of dream recall in patients with epilepsy
2. To describe the characteristics of dreams in epilepsy, the influence of epilepsy on dreams and to characterize the determinants of dream recall frequency in patients with epilepsy We hypothesize that the presence of seizures during sleep will be associated with poorer sleep quality, increased frequency of dream recall, and that we will observe the inclusion of epilepsy symptoms in dream content, particularly in subjects who are aware of their nocturnal seizures and are awakened by them.

ELIGIBILITY:
Inclusion Criteria:

* Patient seen at the epilepsy consultation
* Age 18-65 years
* Certain diagnosis of epilepsy whatever the syndromic diagnosis and the frequency of seizures

Exclusion Criteria:

* major cognitive disorders
* refusal to participate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 consecutives out-patients with epilepsy seen at the consultation of the Epilepsy and Functional Neurology Department, Lyon Neurological Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 347 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2024-01-21 (Actual); Study Completion 2024-01-21 (Actual)

PRIMARY OUTCOMES:
Correlation coefficient between dream recall frequency and nocturnal seizures frequency | Visit 1
  dream recall frequency : question 1 of the EPIDREAM questionnaire nocturnal seizures frequency: question 12 of the EPIDREAM questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Bron, Rhône, France

IPD SHARING:
Plan to Share IPD: No